CLINICAL TRIAL: NCT06320600
Title: Precision Medicine of Diabetes Program in China
Acronym: PDC
Status: Recruiting | Type: Observational
Sponsor: Second Xiangya Hospital of Central South University (Other)
Responsible Party: Principal Investigator, Zhiguang Zhou, director, Second Xiangya Hospital of Central South University
Other Study IDs: PDC
Record Dates: First submitted 2024-02-22; First posted 2024-03-20 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Retrospective PDC cohort: The study will include diabetes patients diagnosed within 1 year (including 1 year) from both inpatient and outpatient medical record systems between January 2022 and December 2022. Each center enrolls approximately 1000 new diabetes patients annually, and it is planned to include 30 centers, with an estimated total of 30,000 participants.
  Interventions: Other: no intervention
- Prospective PDC cohort: The study centers will enroll diabetes patients diagnosed within 1 year (including 1 year) from both outpatient and inpatient services between January 2024 and December 2024. Each center sees approximately 3000 new diabetes patients annually, and it is planned to include 30 centers, with an estimated total of 90,000 participants. The patients will be followed up for a period of 5 years.
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — It's an observational study, no intervention included

SUMMARY:
The prevalence of diabetes has been increasing year by year. According to the International Diabetes Federation (IDF) statistics in 2021, the global number of people with diabetes has reached 537 million. The patient population is large and heterogeneous, and precise diagnosis and treatment of diabetes patients have been a focus of attention. The objective of this study is to clarify the current status of precision classification and diagnosis of diabetes patients through retrospective and prospective cohort studies, and to establish a model for precision classification and diagnosis of diabetes, improving the accuracy of diabetes classification and diagnosis; based on big data of precision medicine for diabetes patients and follow-up cohorts, to establish precise diagnostic, therapeutic, and predictive methods for diabetes; and through multi-omics data analysis, to explore the potential pathogenesis of diabetes, explaining the heterogeneity of patients, and guiding individualized treatment for patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with diabetes according to WHO 1999 criteria

Exclusion Criteria:

* with duration more than 1 year; Diabetes has not been diagnosed by WHO standards in 1999; Absence of medical history data

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The retrospective cohort includes patients diagnosed with diabetes according to WHO 1999 criteria, and the prospective cohort enrolls precisely classified diabetic patients according to "Classification of diabetes mellitus in China: an expert consensus statement".
Sampling Method: Non-Probability Sample
Enrollment: 120000 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
The currency analysis of diabetes classification | July 1st 2023 to December 31th 2023
  To assess the accuracy rate of diabetes classification diagnoses according to "Classification of diabetes mellitus in China: an expert consensus statement" and explore variations across centers in different regions and hospital levels.

SECONDARY OUTCOMES:
To establish a model for predicting diabetic retinopathy | January 1st 2024 to December 31th 2028
  To establish a model for diabetic retinopathy prediction, and calculate the sensitivity and specificity of the model were by comparing with the retinopathy outcome of patients.
To establish a model for predicting diabetic kidney disease | January 1st 2024 to December 31th 2028
  To establish a model for diabetic kidney disease (DKD) prediction, and calculate the sensitivity and specificity of the model were by comparing with the DKD outcome of patients.
To establish a model for predicting diabetic neuropathy | January 1st 2024 to December 31th 2028
  To establish a model for diabetic neuropathy prediction, and calculate the sensitivity and specificity of the model were by comparing with the outcome of patients.

OTHER OUTCOMES:
To establish a model for hypoglycemic therapy | January 1st 2024 to December 31th 2028
  To establish a model for hypoglycemic therapy selection, and compare the rate of HbA1c<7% in patients who are in accordance with the model choice and those who aren't.

CONTACTS AND LOCATIONS:
Locations (1):
- the Second Xiangya Hospital, Changsha, Hunan, China